CLINICAL TRIAL: NCT03714685
Title: A Study in Healthy Subjects Designed to Evaluate the Pharmacokinetic Profile of Firibastat (QGC001) and Active Metabolites Following Administration of Firibastat (QGC001) Prototype Tablet Formulations
Brief Title: Evaluation of the PK Profile of Firibastat Following Administration of Firibastat Prototype Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: QGC001-1QG3; QSC118052 (Other: Quotient Sciences); 2018-001909-89 (EudraCT Number)
Record Dates: First submitted 2018-09-26; First posted 2018-10-22 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Healthy Males
MeSH Terms: interventions — firibastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Firibastat prototype tablet formulations (Experimental): Firibastat (QGC001) 500 mg modified release prototype tablet formulations or immediate release capsule formulation - 1 tablet or 1 capsule administered per period
  Interventions: Drug: Firibastat

INTERVENTIONS:
Drug: Firibastat — Firibastat (QGC001) 500 mg
  Other Names: QGC001

SUMMARY:
This is a single-centre, open-label, non-randomised, period fixed sequence study designed to investigate the PK and safety of Firibastat (QGC001) modified release (MR) prototype tablet formulations and compare this to a reference Firibastat (QGC001) immediate release (IR) capsule formulation in healthy male subjects.

It is planned to enrol 12 subjects to receive single oral doses of investigational medicinal product (IMP).

DETAILED DESCRIPTION:
Subjects will be screened for eligibility to participate in the study up to 28 days before dosing and for each treatment period they will be admitted to the clinical unit on the evening prior to IMP administration (Day -1). On the morning of Day 1, subjects will receive IMP in the fasted state (or following a FDA standard high-fat breakfast, if applicable) and will remain on site until 48 h post-dose. Between the periods, an interim analysis and review of safety and PK data from dosed regimens will be performed in order to determine which Firibastat (QGC001) MR prototype tablet formulation and dose to administer in subsequent periods. A follow-up phone call will take place 7 to 10 days post-final dose to ensure the ongoing wellbeing of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 to 32.0 kg/m2
* Must adhere to the contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* Subjects with pregnant partners
* History of any drug or alcohol abuse in the past 2 years
* Clinically significant abnormal biochemistry, haematology or urinalysis
* Subjects with BP <90/50 mmHg at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profiles of Firibastat (QGC001) and active métabolites of modified release prototype tablet formulations. Assessment of the Maximum Plasma Concentration. | 3 months
  [Cmax]
Pharmacokinetic (PK) profiles of Firibastat (QGC001) and active métabolites of modified release prototype tablet formulations. Assessment of the time at which the Cmax is observed. | 3 months
  [Tmax]
Pharmacokinetic (PK) profiles of Firibastat (QGC001) and active métabolites of modified release prototype tablet formulations. Assessment of the Areas Under the Curve. | 3 months
  [AUC0-24, AUC0-last and AUC0-inf]

SECONDARY OUTCOMES:
Relative bioavailability of Firibastat (QGC001) modified release prototype tablet formulations compared to the immediate release capsule formulation | 3 months
  [AUC0-24 MR / AUC0-24 IR]
Safety and tolerability of single doses of Firibastat (QGC001) by assessing safety haematology and chemistry laboratory tests aggregated as number of patients outside normal ranges. | 3 months
  Basophils, Eosinophils, Haematocrit, Haemoglobin, Lymphocytes, Mean Cell, Haemoglobin, Mean Cell Haemoglobin Concentration, Mean Cell Volume, Monocytes, Neutrophils, Platelet Count, Red Blood Cell Count, White Blood Cell Count
Safety and tolerability of single doses of Firibastat (QGC001) by assessing chemistry laboratory tests aggregated as number of patients outside normal ranges. | 3 months
  Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Bicarbonate, Bilirubin (Total), Calcium, Chloride, Creatine Kinase, Gamma Glutamyl Transferase, Glucose (Fasting), Potassium, Phosphate (Inorganic), Protein (Total), Sodium, Urea
Safety and tolerability of single doses of Firibastat (QGC001) by assessing urinalysis aggregated as number of patients outside normal ranges. | 3 months
  Bilirubin, Blood, Glucose, Ketones, Leukocytes, Nitrites, pH, Protein, Specific gravity, Urobilinogen
Safety and tolerability of single doses of Firibastat (QGC001) by assessing vital signs | 3 months
  Blood pressure (mmHg)
Safety and tolerability of single doses of Firibastat (QGC001) by assessing vital signs | 3 months
  Heart rate (bpm)
Safety and tolerability of single doses of Firibastat (QGC001) by assessing AEs | 3 months
  Adverse events will be recorded from the time of providing written informed consent until discharge from the study at the follow-up visit. During each study visit the subject will be questioned directly regarding the occurrence of any adverse medical event according to the source schedule.
Safety and tolerability of single doses of Firibastat (QGC001) by assessing Twelve-lead ECGs | 3 months
  P wave, T wave, QRS complex, QT interval, RR interval, PR segment, ST segment,

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided